CLINICAL TRIAL: NCT03720821
Title: Cognitive Flexibility Training for Persistent Pain: Neuroimaging Pilot (COFLEX-i)
Acronym: COFLEX-i
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Assistant Professor of Anesthsiology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201808143
Record Dates: First submitted 2018-10-10; First posted 2018-10-25 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain; Knee Pain Chronic; Hip Pain Chronic; Back Pain
MeSH Terms: conditions — Chronic Pain; Back Pain | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Training + fMRI (Experimental): Participants will complete Trail Making Test (TMT) A & B (both electronic and paper-pencil), the paper-pencil Color-Word Matching Stroop Test (CWMST), and its electronic version called "Color Match", and a computer-based subset of NCPT (Neurocognitive Performance Test). In addition, participants will also complete Brief Pain Inventory (BPI), Hospital Anxiety and Depression Scale (HADS), Pain Catastrophizing Scale (PCS), and the Resilience Scale questionnaires at baseline.
  Participants will be provided with the cognitive training module and participants will be required to complete a targeted 36-minute daily training for 35 days.
  Participants will be asked to undergo 2 functional magnetic resonance imaging (fMRI) sessions. One prior to, and one after the 5-week cognitive training period.
  Interventions: Behavioral: Cognitive Training + fMRI

INTERVENTIONS:
Behavioral: Cognitive Training + fMRI — Consented subjects will be asked to participate in the study for up to five months. Patients will be consented at the Washington University Department of Anesthesiology and will be asked to complete baseline resilience, pain, and anxiety and depression questionnaires, along with cognitive tests by pencil and paper that will be administered by a member of the research team. The participants will also be required to complete a computer-based Trails-making test, Color Match test, and NCPT (Neurocognitive Performance Test) battery at baseline, and undergo a functional magnetic resonance imaging (fMRI) session.
  All subjects will be asked to complete the three paper-pencil and computer-based measurements along with repeat pain questionnaire again 1-3 days after completion of training, undergo a second fMRI scan at that time, and complete the questionnaires again 3 months after the completion of training.

SUMMARY:
To determine whether a 5-week computer-based cognitive training intervention results in changes in resting-state functional connectivity (rsFC) within the brain networks.

DETAILED DESCRIPTION:
This project is a single-center prospective pilot study to assess whether cognitive flexibility training through a Lumosity®-based training module over the course a five week timeframe in patients with chronic hip, knee, and back pain results in detectable changes in resting-state functional connectivity (rsFC). The investigators will explore changes in rsFC particularly within the default mode (DMN), frontoparietal (FPN), and cingulo-opercular (CON) brain networks.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 to 70 years old with chronic hip, knee or back pain for >3 months
* Documented moderate to severe chronic pain
* English fluency
* Access to a computer at home and an email account

Exclusion Criteria:

* Lack of email/lack of basic computer skills
* Diagnosed Alzheimer's or documented severe cognitive impairment
* Severely impaired vision or color blindness
* Unable to complete cognitive testing
* An interventional pain procedure within one week prior to enrollment testing
* Scheduled to undergo a pain procedure during the five weeks of cognitive training
* Self-reported claustrophobia
* Contraindication to an MRI scan (i.e. presence of metallic foreign body such as an artificial joint or aneurism clip, implanted pacemaker or spinal cord stimulator)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Changes in resting-state fMRI BOLD signal before and after 5 week cognitive training | 5 weeks
  Changes in resting-state fMRI BOLD (blood oxygenation level dependent) signal before and after 5-week cognitive training, within the default mode, frontoparietal, and cingulo-opercular brain networks.

SECONDARY OUTCOMES:
Association between change in resting-state fMRI BOLD signal and the change in NCPT following cognitive training. | 5 weeks
  Association between change in resting state fMRI BOLD signal and the change in neurocognitive performance test (NCPT) score following 5 weeks of cognitive training.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Background] Haroutiunian S, Nikolajsen L, Finnerup NB, Jensen TS. The neuropathic component in persistent postsurgical pain: a systematic literature review. Pain. 2013 Jan;154(1):95-102. doi: 10.1016/j.pain.2012.09.010. PMID 23273105
- [Background] Smith BH, Torrance N. Epidemiology of neuropathic pain and its impact on quality of life. Curr Pain Headache Rep. 2012 Jun;16(3):191-8. doi: 10.1007/s11916-012-0256-0. PMID 22395856
- [Background] Dworkin RH, Panarites CJ, Armstrong EP, Malone DC, Pham SV. Healthcare utilization in people with postherpetic neuralgia and painful diabetic peripheral neuropathy. J Am Geriatr Soc. 2011 May;59(5):827-36. doi: 10.1111/j.1532-5415.2011.03403.x. PMID 21568954
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Baliki MN, Mansour AR, Baria AT, Apkarian AV. Functional reorganization of the default mode network across chronic pain conditions. PLoS One. 2014 Sep 2;9(9):e106133. doi: 10.1371/journal.pone.0106133. eCollection 2014. PMID 25180885
- [Background] Kucyi A, Salomons TV, Davis KD. Cognitive behavioral training reverses the effect of pain exposure on brain network activity. Pain. 2016 Sep;157(9):1895-1904. doi: 10.1097/j.pain.0000000000000592. PMID 27101426
- [Background] Lamm C, Decety J, Singer T. Meta-analytic evidence for common and distinct neural networks associated with directly experienced pain and empathy for pain. Neuroimage. 2011 Feb 1;54(3):2492-502. doi: 10.1016/j.neuroimage.2010.10.014. Epub 2010 Oct 12. PMID 20946964
- [Background] Vachon-Presseau E, Tetreault P, Petre B, Huang L, Berger SE, Torbey S, Baria AT, Mansour AR, Hashmi JA, Griffith JW, Comasco E, Schnitzer TJ, Baliki MN, Apkarian AV. Corticolimbic anatomical characteristics predetermine risk for chronic pain. Brain. 2016 Jul;139(Pt 7):1958-70. doi: 10.1093/brain/aww100. Epub 2016 May 5. PMID 27190016
- [Background] Bernardy K, Klose P, Busch AJ, Choy EH, Hauser W. Cognitive behavioural therapies for fibromyalgia. Cochrane Database Syst Rev. 2013 Sep 10;2013(9):CD009796. doi: 10.1002/14651858.CD009796.pub2. PMID 24018611
- [Background] Attal N, Masselin-Dubois A, Martinez V, Jayr C, Albi A, Fermanian J, Bouhassira D, Baudic S. Does cognitive functioning predict chronic pain? Results from a prospective surgical cohort. Brain. 2014 Mar;137(Pt 3):904-17. doi: 10.1093/brain/awt354. Epub 2014 Jan 17. PMID 24441173
- [Background] Bowie CR, Harvey PD. Administration and interpretation of the Trail Making Test. Nat Protoc. 2006;1(5):2277-81. doi: 10.1038/nprot.2006.390. PMID 17406468
- [Background] Crowe SF. The differential contribution of mental tracking, cognitive flexibility, visual search, and motor speed to performance on parts A and B of the Trail Making Test. J Clin Psychol. 1998 Aug;54(5):585-91. doi: 10.1002/(sici)1097-4679(199808)54:53.0.co;2-k. PMID 9696108
- [Background] Kortte KB, Horner MD, Windham WK. The trail making test, part B: cognitive flexibility or ability to maintain set? Appl Neuropsychol. 2002;9(2):106-9. doi: 10.1207/S15324826AN0902_5. PMID 12214820
- [Background] Sanchez-Cubillo I, Perianez JA, Adrover-Roig D, Rodriguez-Sanchez JM, Rios-Lago M, Tirapu J, Barcelo F. Construct validity of the Trail Making Test: role of task-switching, working memory, inhibition/interference control, and visuomotor abilities. J Int Neuropsychol Soc. 2009 May;15(3):438-50. doi: 10.1017/S1355617709090626. PMID 19402930
- [Background] Uttl B, Graf P. Color-Word Stroop test performance across the adult life span. J Clin Exp Neuropsychol. 1997 Jun;19(3):405-20. doi: 10.1080/01688639708403869. PMID 9268815
- [Background] Morrison GE, Simone CM, Ng NF, Hardy JL. Reliability and validity of the NeuroCognitive Performance Test, a web-based neuropsychological assessment. Front Psychol. 2015 Nov 3;6:1652. doi: 10.3389/fpsyg.2015.01652. eCollection 2015. PMID 26579035
- [Background] Van Essen DC, Ugurbil K, Auerbach E, Barch D, Behrens TE, Bucholz R, Chang A, Chen L, Corbetta M, Curtiss SW, Della Penna S, Feinberg D, Glasser MF, Harel N, Heath AC, Larson-Prior L, Marcus D, Michalareas G, Moeller S, Oostenveld R, Petersen SE, Prior F, Schlaggar BL, Smith SM, Snyder AZ, Xu J, Yacoub E; WU-Minn HCP Consortium. The Human Connectome Project: a data acquisition perspective. Neuroimage. 2012 Oct 1;62(4):2222-31. doi: 10.1016/j.neuroimage.2012.02.018. Epub 2012 Feb 17. PMID 22366334
- [Background] Glasser MF, Sotiropoulos SN, Wilson JA, Coalson TS, Fischl B, Andersson JL, Xu J, Jbabdi S, Webster M, Polimeni JR, Van Essen DC, Jenkinson M; WU-Minn HCP Consortium. The minimal preprocessing pipelines for the Human Connectome Project. Neuroimage. 2013 Oct 15;80:105-24. doi: 10.1016/j.neuroimage.2013.04.127. Epub 2013 May 11. PMID 23668970
- [Background] Siegel JS, Mitra A, Laumann TO, Seitzman BA, Raichle M, Corbetta M, Snyder AZ. Data Quality Influences Observed Links Between Functional Connectivity and Behavior. Cereb Cortex. 2017 Sep 1;27(9):4492-4502. doi: 10.1093/cercor/bhw253. PMID 27550863
- [Background] Glasser MF, Coalson TS, Robinson EC, Hacker CD, Harwell J, Yacoub E, Ugurbil K, Andersson J, Beckmann CF, Jenkinson M, Smith SM, Van Essen DC. A multi-modal parcellation of human cerebral cortex. Nature. 2016 Aug 11;536(7615):171-178. doi: 10.1038/nature18933. Epub 2016 Jul 20. PMID 27437579
- [Background] Gordon EM, Laumann TO, Adeyemo B, Huckins JF, Kelley WM, Petersen SE. Generation and Evaluation of a Cortical Area Parcellation from Resting-State Correlations. Cereb Cortex. 2016 Jan;26(1):288-303. doi: 10.1093/cercor/bhu239. Epub 2014 Oct 14. PMID 25316338
- [Background] Sporns O, Betzel RF. Modular Brain Networks. Annu Rev Psychol. 2016;67:613-40. doi: 10.1146/annurev-psych-122414-033634. Epub 2015 Sep 21. PMID 26393868
- [Background] Porter S, Torres IJ, Panenka W, Rajwani Z, Fawcett D, Hyder A, Virji-Babul N. Changes in brain-behavior relationships following a 3-month pilot cognitive intervention program for adults with traumatic brain injury. Heliyon. 2017 Aug 4;3(8):e00373. doi: 10.1016/j.heliyon.2017.e00373. eCollection 2017 Aug. PMID 28795168
- [Background] Sandroff BM, Wylie GR, Sutton BP, Johnson CL, DeLuca J, Motl RW. Treadmill walking exercise training and brain function in multiple sclerosis: Preliminary evidence setting the stage for a network-based approach to rehabilitation. Mult Scler J Exp Transl Clin. 2018 Feb 21;4(1):2055217318760641. doi: 10.1177/2055217318760641. eCollection 2018 Jan-Mar. PMID 29497559